CLINICAL TRIAL: NCT07106632
Title: Optimal Personalized Treatment of Early Breast Cancer Using Multi-parameter Analysis: Focus on YOUNGer Women
Brief Title: Optimising Adjuvant Chemotherapy Prescription in Young Patients With Hormone-dependent Breast Cancer Using Genomic Tests
Acronym: OPTIMA-YOUNG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UC-BCG-2409; GA N°101156800 (Other Grant/Funding Number: HORIZON EUROPE); 2024-519655-28-00 (EU CTIS Number); BIG-24-02 (Other: Breast International Group (BIG))
Record Dates: First submitted 2025-06-11; First posted 2025-08-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Early Breast Cancer; Premenopausal Breast Cancer; HR+/HER2- Breast Cancer
Keywords: Adjuvant therapy de-intensification; Care delivery; Quality of Life; Premenopausal Women; Risk stratification
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Drug: In the control arm, the treatment will be as standard of care : chemo-endocrine therapy
- Experimental Arm (Experimental)
  Interventions: Drug: test-directed treatment: allocated treatment will depend on the PAM50 score result (centrally assessed) : chemo-endocrine therapy or endocrine therapy alone

INTERVENTIONS:
Drug: test-directed treatment: allocated treatment will depend on the PAM50 score result (centrally assessed) : chemo-endocrine therapy or endocrine therapy alone — In this experimental arm, the treatment is driven by the score of the Prosigna test. If the score is superior to 60, the patient is considered at hight risk so the patient will receive chemo-endocrine therapy. If the result is under or equal to 60, only endocrine therapy will be prescribed to the patient.
  Arms: Experimental Arm
Drug: In the control arm, the treatment will be as standard of care : chemo-endocrine therapy — Standard treatment: Chemotherapy followed by endocrine therapy
  Arms: Control Arm

SUMMARY:
Rationale:

Around 70 to 80% of breast cancers are so-called "hormone-dependent" (HR+)/HER2-. For more than 50 years, studies have shown that chemotherapy and optimised hormonal treatments (hormone therapy), including a drug associated with ovarian suppression (OFS), improve survival in patients with these cancers, which are characterised by a high risk of relapse. However, younger patients suffer more side effects than older women, particularly from chemotherapy. This can affect their quality of life and reduce their ability to work.

For post-menopausal women, genetic tests exist to assess whether chemotherapy is really necessary in addition to hormonal treatment. However, for high-risk premenopausal patients, chemotherapy is still systematically recommended, as no study has proved that it can be safely avoided. Clinical trials based on risk stratification using genetic tests have not been conclusive, but the majority of premenopausal women included had not received optimal hormone treatment. It is possible that the beneficial effect of chemotherapy is partly due to the artificial menopause it induces. Some experts believe that, for patients with a high clinical risk but a low genetic risk, an optimised hormonal treatment (drug + OFS) could suffice, without the need for chemotherapy.

Objectives:

Main objective: The aim of the study is to determine whether the use of a genetic test (Prosigna®) to decide whether or not to administer chemotherapy produces results as good as standard treatment (systematic chemotherapy) in premenopausal women with hormone-dependent (HR+) breast cancer/HER2-, by assessing their risk of cancer recurrence.

The secondary objectives include verifying whether, in patients with a low Prosigna® score (around 70% of cases), optimised hormonal treatment (including suppression of ovarian function) is as effective as chemotherapy combined with hormonal in treatment preventing cancer recurrence. The study also seeks to compare the efficacy of treatment Prosigna®-guided versus systematic chemotherapy in terms of recurrence and quality of life, as well as economic aspects. Finally, the aim is to understand patients' concerns about the concept of reducing treatment (therapeutic de-escalation) and the way in which this information is communicated to them.

The primary endpoint of the study is to measure the time elapsed between the start of participation in the study and the appearance of an event indicating a return of the cancer. This includes the return of cancer in the same breast or neighbouring areas, the spread of cancer to other parts of the body, the appearance of new cancer in the other breast or death from any cause.

Trial Population:

The study includes women major premenopausal diagnosed with invasive, hormone receptor-positive (ER+) and HER2-negative breast cancer. Patients must have undergone breast and axillary surgery recent and have a tumour sample suitable for analysis by the testProsigna® . They must be able to receive the study treatments Postmenopausal women, women with stage IV breast cancer, women who have already received adjuvant systemic treatment (except short neoadjuvant hormone therapy), women with a recent history of invasive cancer, pregnant women or women who are breast-feeding will not be able to take part in the study.

Interventions:

After agreeing to take part, patients will enter the pre-inclusion period (up to 28 days before randomisation), during which the investigator will carry out all the necessary tests to assess their eligibility. The investigator will then randomise the patients to find out which treatment they have been assigned, no more than 2 weeks later: the experimental group will receive a treatment decided on the basis of the results of a genomic test: either chemotherapy and hormone therapy, or hormone therapy alone. The control group will receive the standard treatment. The treatment and follow-up phases are the same as for standard care. Information on the quality of life patient's will and other information (associated costs, perception of their participation in the study, etc.) also be collected by means of questionnaires completed by the patients during the 5 years following randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent;
2. Female or transgender male persons
3. Age ≥ 35 years
4. Diagnosis of invasive HR-positive (ER≥10% of tumour cells stained positive and any PR expression) HER2-negative (IHC score 0-1+ or 2+ with negative/non-amplified ISH) invasive breast cancer; ER and HER2 determination will be assessed according to latest ASCO/CAP or national guidelines;
5. Breast and axillary surgery completed ≤ 12 weeks from study entry and randomization;
6. Availability of a Formalin-Fixed Paraffin-Embedded (FFPE) tumour sample from surgery to perform Prosigna® analysis.

   Note: in case of receipt of neoadjuvant endocrine therapy the Prosigna® test must be done on the baseline biopsy. Performing the test on the surgical piece or on on-treatment biopsy is not permitted.
7. Tumour size and axillary lymph node status. One of the following must apply:

   1. 1-3 lymph nodes involved AND any invasive tumour size.
   2. node negative (including micrometastases in at least 1 node [i.e. deposit >0.2-2mm diameter]) AND invasive tumour size ≥ 50mm.
8. Multiple ipsilateral breast cancers are permitted provided that at least one tumour meets the tumour size and axillary lymph node entry criteria, and none meet any of the exclusion criteria.
9. Bilateral breast cancers are permitted provided the tumour(s) in one breast meets the eligibility criteria and the other, contralateral tumour is not ER negative and/or HER2 positive and not clinically significant, defined by both of the following:

   1. The contralateral tumour does not fulfil the tumour size and lymph node eligibility criteria required for trial entry; i.e. the following are not acceptable:

      * i. presence of lymph node macro-metastases; .ii. tumour size ≥50mm when there is no lymph node involvement.
   2. The treating physician does not consider that the characteristics of the contralateral tumour alone justify consideration of adjuvant chemotherapy.
10. Fitness to receive adjuvant chemotherapy, as judged by the treating physician;
11. Short term pre-surgical treatment with endocrine therapy, including in combination with non-cytotoxic agents, is allowed providing that the duration of treatment did not exceed 8 weeks;
12. Patients affiliated with or a beneficiary of the local social security system, health social security system, or other local regulatory requirements
13. Patients must agree to use adequate contraception methods for the duration of study treatment and for within 7 months after completing the treatment.

Note : patient with extracapsular nodular transgression are eligible. NOTE: If neoadjuvant endocrine therapy was received, the Prosigna® test must be realized on the baseline biopsy. Performing the test on the surgical specimen or on biopsy taken during treatment is not permitted.

NOTE: Re-excision or complementary mastectomy for close/positive surgical margins should be postponed after chemotherapy completion, if chemotherapy is given; breast reconstruction is allowed after trial entry.

NOTE: The use of approved adjuvant targeted agents (abemaciclib, ribociclib and olaparib) combined to adjuvant endocrine therapy is allowed according to local practice recommendations and availability.

Exclusion Criteria:

* 1. Postmenopausal women. Women who fulfil the following criteria at trial entry will be considered postmenopausal:

  1. Age >45 and natural amenorrhoea of at least 1 year's duration.
  2. Bilateral surgical oophorectomy.
  3. For amenorrhoea not fulfilling the above criteria the diagnosis of postmenopausal status should be supported by hormone measurement: FSH levels must be > 25IU/L with low oestradiol (i.e. within the locally defined postmenopausal range), in the event of doubt measured on 2 occasions preferably 4-6 weeks apart. This applies to women who have undergone hysterectomy without bilateral surgical oophorectomy and are age <60; those ≥60 may be considered postmenopausal.

     NOTE: Hormonal contraception will suppress FSH and oestradiol levels. In those taking oral contraception, levels will recover rapidly on discontinuation. Depo-Provera injectable contraception lasts many months: all women receiving this agent should be considered premenopausal.

     2. Stage IV breast cancer; 3. Start of adjuvant systemic treatment (except for neoadjuvant endocrine therapy for a duration ≤ 8 weeks) before trial entry*; 4. Previous diagnosis of malignancy except:

  <!-- -->

  1. Previous ductal carcinoma in situ (DCIS) or pleomorphic lobular carcinoma in situ (LCIS) of the breast managed by local treatment only;
  2. Previous in situ carcinoma as defined by the International Classification of Diseases for Oncology (ICD-O) including basal cell carcinoma of skin and cervical intraepithelial neoplasia;
  3. Previous invasive malignancy managed by local treatment only AND disease-free for at least 10 years.

     5. Patients enrolled in another therapeutic trial within 30 days of inclusion; 6. Presence of concomitant medical and/or psychiatric comorbidities and/or social problems that might prevent informed consent, treatment compliance or follow up; 7. Person deprived of their liberty or under protective custody or guardianship.

     8. Pregnant women or women who are breast-feeding. 9. Patients unwilling or unable to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures because of geographic, familial, social, or psychological reasons.

     10. Trial entry is dated from of the date the participant signs the consent form or provides remote verbal consent, whichever is earlier.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3380 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-08-15 (Estimated); Study Completion 2038-06-15 (Estimated)

PRIMARY OUTCOMES:
invasive breast cancer free survival (IBCFS) | Time from the date of randomization to the date of the first event (ipsilateral loco-regional invasive breast or distant breast cancer recurrence, contralateral new invasive primary breast cancer or death from any cause), assessed up to 120 months
  Invasive Breast Cancer Free Survival (IBCFS), is defined according to the STEEP version 2.0 system (Tolaney et al., JCO 2021) as the time from the date of randomization to the date of the first event of ipsilateral loco-regional invasive breast cancer recurrence, distant breast cancer recurrence, contralateral new invasive primary breast cancer or death from any cause.

SECONDARY OUTCOMES:
Invasive Breast Cancer Free Survival (IBCFS) in the population with tumours for which the Prosigna® score is below 60 | Time from the date of randomization to the date of the first event (ipsilateral loco-regional invasive breast or distant breast cancer recurrence, contralateral new invasive primary breast cancer or death from any cause), assessed up to 120 months
  Invasive Breast Cancer Free Survival (IBCFS) in the population with tumours for which the Prosigna® score is below the cut-off (≤60) for chemotherapy use, defined according to the STEEP version 2.0 system (Tolaney et al., JCO 2021) as the time from the date of randomization to the date of the first event of ipsilateral loco-regional invasive breast cancer recurrence, distant breast cancer recurrence, contralateral new invasive primary breast cancer or death from any cause.
Distant recurrence free interval (DRFI) | time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer in the global population, assessed up to 120 months
  time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer in the global population
Distant recurrence free survival (DRFS) | time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from any cause in the global population, assessed up to 120 months
  time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from any cause in the global population
Breast cancer specific survival (BCSS) | time from the date of randomization to the date of death from breast cancer in the global population, assessed up to 120 months
  time from the date of randomization to the date of death from breast cancer in the global population
Overall survival (OS) | time from the date of randomization to the date of death from any cause in the global population, assessed up to 120 months
  in the global population, time from the date of randomization to the date of death from any cause in the global population
Distant recurrence free interval (DRFI) in the population with tumours for which the Prosigna® score is ≤60 | time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer assessed up to 120 months
  in the population with tumours for which the Prosigna® score is ≤60 time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer
Distant recurrence free survival (DRFS) in the population with tumours for which the Prosigna® score is ≤60 | time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from any cause, assessed up to 120 months
  in the population with tumours for which the Prosigna® score is ≤60 time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from any cause
Breast cancer specific survival (BCSS) in the population with tumours for which the Prosigna® score is ≤60 | time from the date of randomization to the date of death from breast cancer assessed up to 120 months
  time from the date of randomization to the date of death from breast cancer in the population with tumours for which the Prosigna® score is ≤60
Overall survival (OS) in the population with tumours for which the Prosigna® score is ≤60 | time from the date of randomization to the date of death from any cause assessed up to 120 months
  time from the date of randomization to the date of death from any cause in the population with tumours for which the Prosigna® score is ≤60
Osteoporosis | at ocurrence between baseline and Month 60
  number of non-traumatic fractures
Cardiovascular disease | as ocurrence between baseline and month 60
  major cardioscular events including stroke, myocardial infarction, heart failure and cardiovascular deaths
Fertility | from baseline up to 60 months
  Questions regarding the number of pregnancies, number of living children, any complications during pregnancy or affecting the fetus, as well as the use of contraceptives.
Quality of life (QoL) questionnaire - Core 30 (QLQ-C30) | at baseline, Month 3; Month 6; Month 9; Month 12; Month 24; Month 36; Month 48; Month 60
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR42) | at baseline, month 3, month 6, month 9, month 12, month 24, month 36, month 48, month 60
  this EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR42 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores indicate more severe symptoms or problems for all items.
EQ-ED-5L | at baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
  The EQ-5D-5L (EuroQol 5-Dimension 5-Level) questionnaire is a standardized tool used to assess a person's overall health status. It covers five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from 1 (no problems) to 5 (extreme problems). A patient's health state is summarized by combining their responses into a five-digit code, with each digit representing the level of difficulty in one dimension.
GAD-7 | at baseline, month 6, month 24, month 48, month 60
  The Generalized Anxiety Disorder scale (GAD-7) is a 7-item screening tool used to identify and assess the severity of anxiety disorders. Each item is rated on a 4-point scale: 0 (never), 1 (several days), 2 (more than half the days), and 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating greater anxiety. Based on the total score, individuals are classified into one of four categories: minimal anxiety (0-4), mild anxiety (5-9), moderate anxiety (10-14) or severe anxiety (15-21).
PHQ8 | at baseline, month 6, month 24, month 48, month 60
  The Patient Health Questionnaire-8 (PHQ-8) is an eight-item tool used to screen for and assess the severity of depressive disorders. It focuses on depressive symptoms experienced over the past two weeks. Each item is scored on a scale from 0 (not at all) to 4 (nearly every day), resulting in a total score ranging from 0 to 32. A score of 10 or higher suggests the presence of major depression, while a score of 20 or above indicates severe major depression.
Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) | at baseline, month 6, month 12, month 24, month 36, month 48, month 60
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales: cognitive impairments perceived by the patient (20 items), comments from others (4 items), cognitive abilities perceived by the patient (9 items), and impact on quality of life (4 items). The Perceived Cognitive Impairments and the Comments from Others subscales are rated on 5-point Likerttype scale (from 0 = "Never" to 4 = "Several times a day"). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate perceived cognitive abilities and the impact on quality of life. For all subscales, a higher score represents better cognitive functioning or quality of life.
NCCN Distress thermometer | at baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
  The distress thermometer is an informational tool designed to be shared during appointments to help patients identify their main concerns or side effects and build a personalized action plan. This tool follows a five-step process: patients first rank 3 to 5 top concerns using the NCCN® Distress Thermometer, which contains a simple and reliable 0-to-10 scale for screening distress. In addition, this tool includes a problem list to help users pinpoint sources of distress. It helps patients to reflect on their problems and has proven effective in guiding appropriate psychosocial support and referrals
Return to work | at month 6, month 24, month 36, month 48, month 60
  Questionnaire assessing the support and opportunities available for returning to work after treatment. It also evaluates how treatment and medical appointments impacted work responsibilities during the diagnostic and treatment period, including any changes in remuneration during this time.
Menses and pregnancy status | at baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
  Short question regarding menstrual regularities and pregnancy status.
Fear of Cancer Recurrence (FCRI-SF) | at baseline, month 6, month 24, month 36, month 48, month 60
  A questionnaire regarding the fear of cancer recurrence in the last month. Consisted by 9 items and has been used as a tool to screen for clinical levels of FCR. Each item is rated on a scale from 0 (not at all or never) to 4 (a great deal or several). Higher scores indicate greater FCR severity, with a maximum score of 36.
Motivation to enter the trial (SPECIFIC) | at baseline
  An evaluation designed by The Royal Marsden NHS Foundation Trust to understand patients' experiences in clinical trials and the factors influencing their decision to participate. The questionnaire includes several questions aimed at exploring patients' opinions after enrolling in the trial, as well as the key reasons that motivated their participation.
Recall and expectation on potential treatment related toxicities | at baseline
  Ad hoc questionnaire. Questions about the listed side effects that patients may experience during treatment, as mentioned by the healthcare professional during their medical consultation
Decision Conflict (SURE) | at baseline
  The 4-item SURE screening test is used to evaluate the probability of a patient having decisional conflict. It is composed of four questions (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) and the patient may answer YES or NO. In case of answering at least one "NO", it indicates the probability that a patient experiences clinically significant decisional conflict.
Decision Regret Scale (DRS) | at month 6, month 12, month 36
  This scale measures the distress or remorse after a decision regarding health care. Through 5 different items, in which patients can 1-strongly agree up to 5-strongly disagree a 0-100 scale is formed to evaluate the patient satisfaction of the decision taken.
Physical Activity Levels (IPAQ) | at baseline, month 6, month 12, month 24, month 48, month 60
  A questionnaire regarding the physical activities in the last 7 days. In the short form of the IPAQ questionnaire 7 questions are made regarding the intensity of physical activity. The results are converted into METs, a method to quantify energy spent in physical activities. Based on this, 3 different levels are proposed: low, moderate or high.
Body Mass Index | at baseline, month 6, month 12, month 24, month 48, month 60
  Body Mass Index (BMI) is a widely used measure to assess whether an individual's weight is appropriate for their height. It is calculated using the formula: BMI = weight (kg) / height (m²). Based on the resulting value, BMI is categorized as follows: Underweight: BMI < 18.5; Normal weight: BMI 18.5 - 24.9; Overweight: BMI 25.0 - 29.9; Obesity: BMI ≥ 30.0
Tobacco and alcohol consumption | at baseline, month 6, month 24, month 48, month 60
  Assessment includes the frequency of alcohol consumption in the last 12 months and smoking status of the patient, including the quantity consumed in both cases.
Self-reported adherence to ET (VOILS) | at month 6, month 12, month 18, month 24, month 30, month 36, month 42, month 48, month 54, month 60
  The self-reported adherence questionnaire aims to assess how often patients forget to take their hormone therapy and to identify the reasons behind missed doses.
Use of Healthcare Resources | at baseline, month 6, month 24, month 36, month 48, month 60
  Questionnaire that aims to list different aspects of healthcare services usage in the previous 3 months: inpatient stay, outpatient consultation, number and type of exams done. There are also questions regarding the amount spent for travels to attend hospital or other health and social care appointments, including any unplanned visits.
Score of perceived ease of use (SUS) | at month 3
  The System Usability Scale (SUS) is a standardized survey designed to evaluate the perceived usability of a system or product. It generates a score ranging from 0 to 100, with higher scores indicating better usability. The SUS consists of 10 statements, each rated on a 5-point Likert scale, where 1 means "strongly disagree" and 5 means "strongly agree." Respondents' answers reflect their overall satisfaction and ease of use of the system.
Distant recurrence free interval (DRFI) | time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer in the global population, assessed up to 12 months
  time from the date of randomization to the date of the first event of distant recurrence of breast cancer or death from breast cancer in the global population

CONTACTS AND LOCATIONS:
Overall Officials: Ines Vaz-Luis, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: Undecided